CLINICAL TRIAL: NCT05941377
Title: Enhanced Versus Standard Blood Pressure Lowering on Intracranial Aneurysm Rupture or Growth
Brief Title: China Antihypertensive Trial for Intracranial Aneurysm (ChATIA-1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: RenJi Hospital (Other); Guangzhou Red Cross Hospital (Other); Jiangnan University Medical Center (Unknown); Binzhou Medical University (Other); Beijing Friendship Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2023-050-01
Record Dates: First submitted 2023-06-29; First posted 2023-07-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Unruptured Intracranial Aneurysm
Keywords: Unruptured Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard blood pressure lowering (SBPL) group (Experimental)
  Interventions: Other: blood pressure lowering
- enhanced blood pressure lowering (EBPL) group (Experimental)
  Interventions: Other: blood pressure lowering

INTERVENTIONS:
Other: blood pressure lowering — For EBPL group, patients are required to keep blood pressure at 100-120 mmHg. For SBPL group, patients are required to keep blood pressure at 120-140 mmHg.

SUMMARY:
The goal of this randomized controlled trial is to evaluate the benefits and safety of controlled hypotension in Chinese patients with unruptured intracranial aneurysms(UIA).

The main questions it aims to answer are:

* To provide high-level evidence of the benefits and safety of controlled hypotension in patients with UIA.
* To provide evidence-based medical evidence for blood pressure control of patients with UIA in neurosurgery, and promote the progress of accurate individual management of patients. In this study, the main intervention is enhanced blood pressure lowering in patients with UIA.

All Patients will be randomly assigned to either the standard blood pressure lowering (SBPL) group or the enhanced blood pressure lowering (EBPL) group.

ELIGIBILITY:
Inclusion criteria

1. Age 18-75.
2. Chinese ethnicity.
3. Unruptured saccular intracranial aneurysm (UIA) identified by computational tomography angiography, magnetic resonance angiography or digital subtraction angiography.

   1. Maximal size of UIA at largest dimension < 7 mm
   2. The morphology of UIA is regular (no bleb(s) or secondary aneurysm(s) protruding from the UIA fundus or bi-/ multi-lobular UIA fundus)
   3. UIA receiving conservative treatment
4. History of primary hypertension (as diagnosed per standard of care)
5. Systolic blood pressure (SBP) on 2 consecutive visits:

   SBP: 130-180 mmHg on 0 or 1 antihypertensive medication. SBP: 130-170 mmHg on up to 2 antihypertensive medications. SBP: 130-160 mmHg on up to 3 antihypertensive medications. SBP: 130-150 mmHg on up to 4 antihypertensive medications
6. Good medication adherence (Morisky Medication Adherence Scale ≥6)
7. Obtain informed consent from patient or legal representative

Exclusion criteria:

1. Patients with neurological symptom related to UIA, such as sentinel headache, oculomotor paralysis and so on.
2. Patients with additional active intracranial disease including vasculopathy, arteriovenous malformation/fistula, cancer, traumatic brain injury etc.
3. Patients with fusiform, dissecting, blister, traumatic, mycotic/ bacterial, myxomatous, and tumor-associated UIAs are excluded.
4. Patients with history of polycystic kidney disease, rheumatic disease or autoimmune disease.
5. Patients with family history of intracranial aneurysm (defined when two direct relatives of patients within three generations have intracranial aneurysms or aneurysmal subarachnoid hemorrhage).
6. Patients with known secondary cause of hypertension.
7. Patients with myocardial infarction, ischemic stroke, symptomatic heart failure during the past 3 months.
8. Patients with a medical condition likely to limit survival to less than 2 years.
9. Patients during pregnancy and perinatal period.
10. Any concurrent serious illness that would interfere with the outcome assessments including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease.
11. Inability or unwillingness of patient or legal representative to give written informed consent.
12. Participation in a concurrent interventional medical investigation or clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
UIA instability | 24 months
  The primary outcome is UIA instability (rupture, growth on radiological examination, or occurrence of aneurysm-related symptoms [sentinel headache and oculomotor paralysis]).
safety endpoint | 24 months
  The safety endpoint is any ischemic cerebral or cardiac events. This includes one or more of the following: new or more frequent transient ischemic attack, new clinical or radiological ischemic stroke, angina, new myocardial infarction, or reperfusion therapy for myocardial infarction.

SECONDARY OUTCOMES:
UIA rupture events | In 24 months
  UIA rupture events in 24 months
UIA growth events | In 24 months
  UIA growth events in 24 months
Change in average Wall Enhancement Index | At baseline and 24th month
  Change in average Wall Enhancement Index (WEI) at baseline and 24th month

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zheng K, Mo S, Wen Z, Li J, Miao Z, Lu X, He H, Cao Y, Zhao B, Levitt MR, Chen L, Wang S, Zhu C, Liu Q. Enhanced versus standard blood pressure lowering on intracranial aneurysm rupture or growth (ChATIA-1 trial): protocol for a multi-centered, prospective, open-label randomized controlled trial. Front Neurol. 2026 Jan 7;16:1627936. doi: 10.3389/fneur.2025.1627936. eCollection 2025. PMID 41573399